CLINICAL TRIAL: NCT06529211
Title: Effect of Ultrasound Cavitation Versus Whole Body Vibration on Abdominal Fat in Obese Adolescent Females: a Randomized Controlled Trial
Brief Title: Effect of Ultrasound Cavitation Versus Whole Body Vibration on Abdominal Fat in Obese Adolescent Females
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Christina Samir Harmakes, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004858
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Abdominal Obesity
MeSH Terms: conditions — Obesity, Abdominal | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low caloric diet group (Active Comparator): low-caloric diet of 1500 kcal/day.
  Interventions: Dietary Supplement: Low caloric diet
- ultrasound cavitation group (Experimental): The participants will be treated by ultrasound cavitation, in addition to the low-caloric diet of 1500 kcal/day.
  Interventions: Dietary Supplement: Low caloric diet; Device: Ultrasound cavitation
- whole-body vibration group (Experimental): The participants will be treated by whole body vibration, in addition to the low-caloric diet of 1500 kcal/day.
  Interventions: Dietary Supplement: Low caloric diet; Device: Whole body vibration

INTERVENTIONS:
Dietary Supplement: Low caloric diet — Low caloric diet: the participants will receive low caloric diet program (1500 Kcal/ day) for 6 weeks as follows: 45% carbohydrate, 20% fat and 35% proteins of total calorie intake.
Device: Ultrasound cavitation — Ultrasound cavitation + Low caloric diet Low caloric diet program (1500 Kcal/ day): for 6 weeks.
  Ultrasound cavitation: It will be on abdomen for 30 minutes/session, 2 sessions/week for 6 weeks as follows:
  * The participants will be in supine lying position and the abdomen is divided into two sides right and left from the midline.
  * The Ultrasound pulsed waves will be set with power input (AC100/ 240V), frequency (40 KHz), and Power output (45W). This will be for 15 minutes on each abdominal side.
  Arms: ultrasound cavitation group
Device: Whole body vibration — Whole body vibration + Low caloric diet Low caloric diet program (1500 Kcal/ day) for 6 weeks.
  Whole body vibration: for 30 minutes/session, 2 sessions/week for 6 weeks as follows:
  * The participants will begin with a brief warm-up for 5 minutes by doing deep breathing exercises.
  * Then they will stand with feet shoulder-width apart on the platform while holding handrails to maintain balance and stability. They will be instructed to relax and allow the vibrations to pass through her body. This will be applied for 20 minutes per session.
  * The vibration will be started with lower settings and gradually will be increased till the desired frequency and amplitude (45 HZ) will be reached.
  * After the session will be completed, the participant will be instructed to cool down gradually by doing deep breathing for 5 minutes to help their body to return to a resting state. They will be advised to drink plenty of water to be hydrated and recovered after the WBV session.
  Arms: whole-body vibration group

SUMMARY:
This study aims to determine the differences between the effect of ultrasound cavitation and whole-body vibration on abdominal fat in obese adolescent females

DETAILED DESCRIPTION:
Adolescence is a critical time associated with the development of obesity. About 80% of adolescents with obesity will continue to have this condition as an adult.

Obesity during adolescence is associated with a number of short- and long-term diseases including hypertension, diabetes mellitus type 2, hyperlipidemia, obstructive sleep apnea, psychological distress and future cardiovascular complications.

The investigators showed that there is an increasing demand for non-surgical procedures in the management of obesity that led to the development of non-invasive techniques for reducing localized subcutaneous adipose tissue.

One of these techniques is focused ultrasound cavitation. Research studies showed some benefits in the treatment of excess abdominal fat deposits with reduction in fat circumference without significant side effects.

Also, another non-invasive technique is whole body vibration (WBV). Some studies showed that when it is combined with dietary intervention leads to body weight reduction and improvement of overall body composition and fat reduction including abdominal fat

Both ultrasound cavitation (UC) and whole-body vibration (WBV) are non-invasive modalities with many positive effects on abdominal fat in obese adolescent females. The effect of both the UC and WBV has been separately investigated in previous studies. Though, no studies were found to compare the effect of both modalities in the management of abdominal fat in obese adolescent females. Therefore, this study will be conducted to explore the effect of UC versus WBV on abdominal fat in obese adolescent females.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent females suffer from abdominal obesity.
* Their ages will be ranged from 17 to 25 years old.
* Their body mass index (BMI) will be ranged from 30 to 35 kg/m2.
* Their waist circumference will be > 88 cm.
* Their WHR will be more than 0.88.

Exclusion Criteria:

Females will be excluded from the study if they have:

* Thyroid, hepatic and kidney disorders.
* Diabetes mellitus, coronary artery diseases, hypertension and congestive heart failure.
* Recent abdominal surgical scar or umbilical hernia.
* History of orthopedic implants insertion or cardiac pacemaker implantation.

Ages: 17 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Adolescent females
Enrollment: 60 (Estimated)
Dates: Start 2024-07-22 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Weight | Within 6 weeks
BMI | Within 6 weeks
  Weight/ height scale will be used to measure the weight and height of all females in all groups to calculate their BMI before and after treatment according to the following equation BMI = weight/ height² (kg/m²)
Waist circumference | Within 6 weeks
  It is a measurement taken around the waist at the level of the narrowest part of the torso, typically located between the bottom of the rib cage and the top of the hip bones (iliac crest). It is used as an indicator of central obesity. However, as a general guideline, a waist circumference of over 35 inches (88 cm) in women is often considered high and indicative of an increased health risk .
Waist to hip ratio (WHR) | Within 6 weeks
  Waist-to-hip ratio (WHR) is a measurement that compares the circumference of the waist to that of the hips. The waist circumference is measured at the narrowest point of the torso, usually just above the belly button (umbilicus), and the hip circumference is measured at the widest part, 9 around the buttocks at level of greater trochanters; then dividing the waist circumference by the hip circumference. The formula is as follows: WHR = Waist Circumference / Hip Circumference. For women, a WHR above 0.85 is often considered high and indicative of an increased health risk.
Abdominal skinfold thickness | Within 6 weeks
  Abdominal skinfold thickness is a specific measurement used to estimate the amount of subcutaneous fat in that area. It provides insights into the distribution of fat in the abdominal region. The measurement is typically taken at a site approximately 2 cm to the right side of the belly button, and the skinfold is pinched with calipers to measure the thickness. The measurement process involves firmly grasping the skin and underlying fat tissue with the calipers, ensuring that only the skin and fat are included in the measurement and not muscle or other tissues. The measurement is recorded in millimeters (mm)
Bioelectrical impedance analysis (BIA) | Within 6 weeks
  In BIA, a small, safe electrical current is passed through the body using electrodes typically placed on the hands and feet. The electrical current encounters resistance from tissues with lower water content, such as fat and bone, while it easily passes through tissues with higher water content, such as muscle. By measuring the impedance (resistance and reactance) of the electrical current, BIA devices can estimate body composition parameters such as body fat percentage, lean body mass, and hydration levels. BIA can provide a quick and non-invasive estimation of body composition. Also, it is a useful tool for tracking changes in body composition over time and monitoring progress in fitness or weight loss programs.

CONTACTS AND LOCATIONS:
Overall Officials: Azza Kassab, Study Chair — Cairo University; Manal El-Shafei, Study Director — Cairo University; Mohamed AboEleinen, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol